CLINICAL TRIAL: NCT04748874
Title: Immediate Versus Postponed Single Blastocyst Transfer in Modified Natural Cycle Frozen Embryo Transfer (mNC-FET): a Multicenter Randomized Controlled Trial
Brief Title: Immediate Versus Postponed Single Blastocyst Transfer in mNC-FET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kristine Loessl, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-19086300
Record Dates: First submitted 2020-12-18; First posted 2021-02-10 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Infertility; IVF
Keywords: Frozen embryo transfer; Immediate FET; Postponed FET; mNC FET
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate mNC-FET (Experimental): In the immediate arm, patients undergo mNC-FET in the menstrual cycle immediately following oocyte retrieval and failed fresh embryo transfer or freeze-all.
  Interventions: Procedure: Immediate mNC-FET
- Postponed mNC-FET (No Intervention): Standard procedure where mNC-FET is performed at least one full menstrual cycle after failed fresh embryo transfer or freeze-all cycle.

INTERVENTIONS:
Procedure: Immediate mNC-FET — In the immediate arm, patients undergo mNC-FET in the menstrual cycle immediately following oocyte retrieval and failed fresh embryo transfer or freeze-all.
  Arms: Immediate mNC-FET

SUMMARY:
The purpose of this randomized controlled trial is to investigate if immediate single blastocyst transfer (in the first menstrual cycle following oocyte retrieval) is non-inferior to standard postponed single blastocyst transfer (in the second or subsequent menstrual cycle following oocyte retrieval) in modified natural cycle frozen-thawed embryo transfer (mNC-FET) in terms of live birth rate.

DETAILED DESCRIPTION:
The study is a multicenter randomized non-blinded controlled trial with the purpose of investigating if immediate mNC-FET is non-inferior to standard postponed mNC-FET in terms of live birth rate and other obstetric- and neonatal outcome.

Several fertility clinics in Denmark will participate in the recruitment of patients. All clinics perform standardized treatments according to the public health care system in Denmark. Patient enrolment is expected to begin in February 2021 and continue until December 2024.

The study population will consist of 464 patients undergoing mNC-FET after a fresh IVF/ICSI cycle that did not result in a viable pregnancy, or after a freeze-all cycle. Eligible patients will be recruited if they fulfil the inclusion criteria and none of the exclusion criteria. Patients will be randomized 1:1 by simple randomization to one of the following study arms:

I. Immediate mNC-FET In the Immediate arm, patients will undergo mNC-FET in the menstrual cycle immediately following oocyte retrieval with failed fresh embryo transfer or freeze-all.

II. Postponed mNC-FET In the Postponed arm, mNC-FET is performed at least one full menstrual cycle after the fresh embryo transfer or freeze-all cycle, which means that the first FET following the fresh cycle is not started until the second menstrual bleeding or later.

Patients who did not conceive after fresh embryo transfer, or patients undergoing a freeze-all cycle, will be invited to participate in the study if they have at least one vitrified blastocyst with embryo quality of minimum 3BB according to the Gardner score.

Patient related data and blood samples will be collected at baseline, day of ovulation trigger, day of blastocyst transfer and day of pregnancy testing for all participants. Patients enrolled at Rigshospitalet will have additional blood samples collected in the early- and mid-luteal phase. LH, FSH, progesterone and estradiol will be measured at all time-points. Blood used for these consecutive analyses will be destroyed immediately as a part of the daily laboratory routine. Additional blood samples will be collected and kept in a biobank at Rigshospitalet if patients agree. Patients are asked to sign a separate informed consent form for storage of blood samples in a biobank for future research projects.

Quality of life questionnaires will be collected at baseline and in the mid-luteal phase. If the woman has a partner, her or she will be asked to fill out quality of life questionnaires at the same time-points (requires separate informed consent).

Transvaginal ultrasound scans (TVUS) will be performed at baseline (cycle day 2-5) and on the day of ovulation trigger. Ovulation trigger by hCG (6500 IU) is administered when the dominant follicle reaches 17-18 mm. Single blastocyst warming and ultrasound guided transfer is performed 6 days after hCG trigger. If the patient conceives, a transvaginal scan will be performed at 7-8 weeks of gestation in order to assess viability and crown-rump length.

To compare ovarian morphology of the first cycle immediately following oocyte retrieval to the standard postponed cycle, a number of parameters, including ovarian volume and size and appearance of follicular structures >10 mm, will be assessed with 2- and 3D TVUS at baseline and the day of hCG-trigger. 2D scans will be performed for all participants. 3D scans will be performed on a subgroup of participants at the same time points.

In case of pregnancy and delivery, data will be collected from the patient's medical records as well as the new-born child's birth records for registration of obstetric and neonatal outcomes. The custodians will be asked permission to access the upcoming child's journal for the purpose of gathering information about the birth and health of the child within the first year of life.

Data will be transferred to an online eCRF; REDCap. The REDCap database has a complete audit trail and is based on anonymous subject identification numbers used in the trial. Data are backed up daily and stored on a server located in a locked facility in Denmark.

The study is designed as a non-inferiority trial. A non-inferiority margin of 10% is considered clinically relevant. We expect a LBR of 25% per randomized study participant after postponed single blastocyst transfer in mNC-FET, which is considered the standard treatment. If there is truly no difference between the standard- and intervention treatment 464 participants (n=232 in each group) are required to be 80% sure that the upper limit of a one-sided 95% confidence interval (CI) (or equivalently a 90% two-sided CI) will exclude a difference in favour of the standard group of more than 10%.

As primary outcome, difference in LBR will be evaluated by means of risk difference with one-sided 95% CI. Non-inferiority will be concluded if the CI excludes a difference of more than 10% in favour of the standard treatment in intention-to-treat (ITT) and per protocol (PP) analyses. Difference in LBR per-transfer will be assessed as a secondary outcome by risk difference with 95% CI. Rate of positive hCG, ongoing pregnancy, miscarriage and cancelled cycles will be assessed by risk differences with 95% CI in PP, ITT and per-transfer analyses as outlined for LBR. Mean day of ovulation and mean levels of hormones will be compared with T-test. Hormone levels known to have a skewed distribution will be log-transformed prior to analysis. Number of ovarian follicular structures >10 mm will be assessed with a chi-squared-test in a PP analysis. Time-to-pregnancy and live-birth per delivery will be compared in Kaplan-Meier plots and using log-rank test. Rates of pregnancy-related complications and adverse neonatal outcomes per delivery will be assessed using Fisher's exact test. Data on quality of life and psychosocial status will be obtained in a validated self-reported survey expressed by Likert based 5-scale items and compared by non-parametric Mann-Whitney U-tests. Statistical analyses will be performed using R.

Numbers and reasons for drop-out and cancellation will be tabulated for the two treatment groups and descriptive tables will be compiled for comparison of characteristics of drop-outs, cancelled cycles and completers within and between the groups. We anticipate a drop-out rate of at most 5% and a cancellation rate of at most 5%. In case of a differential or larger than expected drop-out or cancellation rate, potential biases will be discussed along with any discrepancies between the results of the PP, ITT and per-transfer analyses and conclusions will be drawn accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for FET in a modified natural cycle
* Regular menstrual cycle (23-35 days)
* Vitrified day 5 or 6 blastocyst
* Blastocyst Gardner score > or = 3BB at the day of vitrification

Exclusion Criteria:

* Uterine malformations or presence of hydrosalpinx
* Submucosal uterine myomas
* Uterine polyps
* Allergy to standard fertility medication
* Contradiction to standard fertility medication
* Male of female HIV, hepatitis B or C
* Preimplantation Genetic Testing (PGT) in the fresh cycle
* Severe OHSS during the fresh cycle (defined as need for ascites drainage and/or hospital admission)
* Oocyte donation
* Testicular sperm aspiration (TESA)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 464 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Live birth rate per randomized patient | One-year follow-up after a positive pregnancy test
  Live birth rate in patients randomized to immediate versus postponed FET
Live birth rate per protocol | One-year follow-up after a positive pregnancy test
  Live birth rate in patients randomized to immediate versus postponed FET minus dropouts

SECONDARY OUTCOMES:
Live birth rate per blastocyst transfer | One-year follow-up after a positive pregnancy test
  Live birth rate in patients receiving blastocyst transfer in the immediate versus postponed arm
Positive hCG rate per randomized patient and per blastocyst transfer | 16 days after ovulation trigger (hCG+16)
  Rate of positive hCG in the immediate versus postponed arm
Ongoing pregnancy rate per randomized patient and per blastocyst transfer | Ultrasound at 7-8 weeks of gestation
  Ongoing pregnancy rate (visualisation of an intrauterine gestational sac containing a foetus with heartbeat) in the immediate versus postponed arm
Biochemical pregnancy loss | 16 days after ovulation trigger (hCG+16) and up to 7-8 weeks
  Rate of biochemical pregnancy loss (positive hCG spontaneously declining before visualization of an ongoing pregnancy) in the immediate versus postponed arm
Clinical pregnancy loss | Routine ultrasound at 7-8 weeks of gestation or ad hoc ultrasound before 22 weeks of gestation
  Rate of clinical pregnancy loss (clinically recognised pregnancy that is lost before 22+0 weeks of gestation) in the immediate versus postponed arm
Cycle cancellation | 16 days after ovulation trigger (hCG+16) and through study completion, up to 1 year
  Cycle cancellation rate in the immediate versus postponed arm
Reason for cycle cancellation | 16 days after ovulation trigger (hCG+16) and through study completion, up to 1 year
  Reason for cycle cancellation in the immediate versus postponed arm
Number of ovarian follicular structures >10 mm | At baseline and on day of ovulation trigger (hCG+0), up to 1 month
  Number of ovarian follicular structures >10 mm in the immediate versus postponed arm
Day of ovulation | From first day of FET cycle to the day of ovulation trigger (hCG+0), up to 1 month
  Day of ovulation in the immediate versus postponed arm
Endocrinology of the luteal phase | Baseline, day of ovulation trigger (hCG+0), early luteal phase* (hCG+4), day of transfer (hCG+6) and mid-luteal phase* (hCG+11)(*only at Rigshospitalet), within one FET cycle, up to approximately 1 month
  Hormone levels in blood in the immediate versus postponed arm
Time-to-pregnancy | From day of ovarian stimulation to day of clinical pregnancy, up to 1 year
  Time-to-pregnancy in the immediate versus postponed arm
Time-to-live-birth | From day of ovarian stimulation through study completion, up to 18 months
  Time-to-live-birth in the immediate versus postponed arm
Pregnancy related complications | One-year follow-up after a positive pregnancy test
  Pregnancy related complications in patients receiving immediate versus postponed FET
Neonatal outcome | One-year follow-up after a positive pregnancy test
  Neonatal outcome in children of patients in patients receiving immediate versus postponed FET
Quality of life assessment | Baseline and mid-luteal phase (hCG+11), up to 1 month
  Quality of life in the immediate versus postponed arm, questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anja B Pinborg, Prof. DMSc, Study Director — Fertility department , Rigshospitalet
Locations (1):
- Fertility department, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data from the trial will be shared according to the ICJME guidelines. On request, data can be shared with parties presenting relevant aims for the use of data. Purposes and financial aspects of the other party must be approved by the steering committee of the "FET-immediate" research team. Data will not be shared with groups presenting research projects with the same aims or purposes as ours. No data will be shared until three months after publication of papers reporting the primary and secondary outcomes of the trial. Any new research project must be approved by Danish authorities. The requesting party will cover the costs for data sharing.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Bergenheim S, Saupstad M, Colombo C, Moller JE, Bogstad JW, Freiesleben NC, Behrendt-Moller I, Praetorius L, Oxlund B, Nohr B, Husth M, Lokkegaard E, Sopa N, Pinborg A, Lossl K, Schmidt L. Psychosocial and physical wellbeing in women and male partners undergoing immediate versus postponed modified natural cycle frozen embryo transfer after ovarian stimulation and oocyte pick-up: a sub-study of a randomized controlled trial. Hum Reprod. 2025 Jan 1;40(1):96-109. doi: 10.1093/humrep/deae260. PMID 39673443
- [Derived] Bergenheim SJ, Saupstad M, Pistoljevic N, Lyng Forman J, Larsen EC, Bogstad JW, Fynbo M, Hashem N, Freiesleben NC, Nohr B, Andersen LF, Humaidan P, Ziebe S, Pinborg AB, Lossl K. Immediate versus postponed single blastocyst transfer in modified natural cycle frozen embryo transfer (mNC-FET): a study protocol for a multicentre randomised controlled trial. BMJ Open. 2021 Oct 27;11(10):e053234. doi: 10.1136/bmjopen-2021-053234. PMID 34706963